CLINICAL TRIAL: NCT06967922
Title: Evaluation of Analytic-integrative Cognitive Behavioural Therapy for Acute Insomnia Disorder (Stress)
Brief Title: Impact of Analytic-integrative Cognitive Behavioural Therapy on Acute Insomnia Disorder (Stress)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICBT for AID
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Acute Insomnia Disorder
Keywords: Acute insomnia disorder; Analytic-Integrative Cognitive Behavioural Therapy; stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance analysis - integrated cognitive behavioral therapy (Experimental)
  Interventions: Behavioral: Analytic-Integrative Cognitive Behavioural Therapy
- Receive sleep hygiene education (Active Comparator)
  Interventions: Other: Sleep hygiene education

INTERVENTIONS:
Behavioral: Analytic-Integrative Cognitive Behavioural Therapy — Analytic-Integrative Cognitive-Behavioural Approach: Initial Interview for Information Gathering: comprehensive collection of patient information; Assessment: collection of multidimensional factors; Diagnosis: insomnia and co-morbidities; Analytic-Integrative Analysis for Treatment Decision Making.
  Arms: Acceptance analysis - integrated cognitive behavioral therapy
Other: Sleep hygiene education — Participants will receive Sleep Hygiene Education (SHE) alone for 6 weeks. SHE involves education on maintaining consistent sleep schedules, creating a sleep-conducive environment, reducing stimulant use (e.g., caffeine, alcohol), and promoting healthy daily routines to improve sleep quality.
  Arms: Receive sleep hygiene education

SUMMARY:
The main objective of this study, conducted in a population with acute insomnia disorder (stress), was to investigate the efficacy of Analytic-Integrative Cognitive Behavioural Therapy in the treatment of acute insomnia disorder (stress).

DETAILED DESCRIPTION:
Acute insomnia disorder, also known as short-term insomnia disorder, is basically characterised by difficulties with short-term sleep onset and maintenance and results in feelings of sleep dissatisfaction. When insomnia arises in response to a stressful life event (painful loss of a loved one, major illness, or divorce), associated features may include anxiety, worry, sadness, or depression related to the specific stressor. Medications are a common form of treatment for acute insomnia disorders, and while they may improve the patient's clinical symptoms, the overall results are not very satisfactory. Cognitive behavioural therapy, as a non-pharmacological treatment, has become the first-line recommended solution in the insomnia treatment guidelines of China and the United States, which can correct patients' wrong sleep cognition and bad sleep habits, establish correct sleep-wake cognition, and also improve mental health. Compared with sedative-hypnotic medications, it has no adverse reactions and does not affect daytime function, making it a green and safe treatment method. Based on the exact efficacy of cognitive behavioural therapy in improving insomnia, and also considering the diverse causes of acute insomnia disorder (stress), we analyse-integrate the analysis of the patient's specific situation, and we propose to treat acute insomnia disorder through analytical-integrative cognitive behavioural therapy, formulate an individualized treatment plan to improve the therapeutic effect, and prevent the patient from developing in the direction of chronic insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. meeting the DSM-5 diagnostic criteria for insomnia disorder;
2. a total score of >5 on the Pittsburgh Sleep Quality Index (PSQI);
3. age ≥18 years old, with junior high school education or above;
4. voluntarily participating in this study and signing an informed consent form;
5. the diagnostic criteria for acute insomnia disorder (duration of the disease less than 3 months).

Exclusion Criteria:

1. people with comorbid serious physical or severe mental illnesses, suicide risk;
2. clinically diagnosed or suspected sleep breathing disorder, restless legs syndrome and sleep-wake rhythm disorder, shift workers;
3. pregnant and breastfeeding women;
4. people who are currently undergoing any psychological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The change of Pittsburgh Sleep Quality Index (PSQI) total scores from baseline to 6 weeks. | Baseline, 6 weeks
  The PSQI consists of 7 factors ranging from 0 to 3 points, and the total score ranges from 0 to 21 with higher scores indicating poorer quality.

SECONDARY OUTCOMES:
The change of Beck Depression Inventory (BDI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BDI assessing the existence and severity of symptoms of depression consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe depressive symptoms.
The change of Beck Anxiety Inventory (BAI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BAI assessing the existence and severity of symptoms of anxiety consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe anxiety.
The change of Snaith-Hamilton Pleasure Scale (SHAPS) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The SHAPS assessing anhedonia consists of 14 items, and the total score ranges from 14 to 56 with higher scores indicating more serious the anhedonia.
The change of Insomnia severity index (ISI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The ISI reporting insomnia symptoms severity consists of 7-items on a 5-point Likert scale, and the total score ranges from 0 to 28 with higher scores indicating more severe insomnia.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No